CLINICAL TRIAL: NCT07021274
Title: DBT Skill Training for Autistic Adults With Difficulties in Emotion Regulation: a Feasibility Study.
Brief Title: DBT Skill Training for Autistic Adults With Difficulties in Emotion Regulation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: The Dam Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 836937
Record Dates: First submitted 2025-05-19; First posted 2025-06-13 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Difficulties of Emotion Regulation; Self-harm Behavior; Autism Spectrum Disorder
Keywords: Autisim; emotion regulation; DBT skills training; adults; ASD; Feasibility; Autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study is a mixed-method feasibility study without a control group. With measurements pre and post treatment intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participate in DBT skills training (Experimental): The intervention period will be from August 2025- February 2027.
  DBT- skills is a group skills training component of Dialectical Behaviour therapy a comprehensive treatment focused on extensive difficulties in emotion regulation. In this project, the investigators will use the standard DBT skill-training model with an addition of Autism specific interventions and adjustments.
  The DBT-SUD Skills intervention consists of:
  2-3 sessions with a DBT therapist focusing on treatment orientation - mapping the patients' goals, obstacles, and resources, DBT- hierarchy, and commitment.
  Skills training - 28, two-hour sessions - once a week.
  1 status and evaluation session half-way through the skills training.
  1 summary session with a focus on goals reached and troubleshooting.
  Two DBT therapists lead the group, and each group consists of approx. 4-6 participants.
  Interventions: Behavioral: DBT skills training adjusted to autistic needs

INTERVENTIONS:
Behavioral: DBT skills training adjusted to autistic needs — Adjustments to fit the specific learning style of people with autism. Simplified skills - fewer words, ,more pictures, autism relevant examples. Hands- on training using props and role play. adjustments so sensory sensitivities.

SUMMARY:
One in 44 has autism, 70% of them have additional mental health challenges. Currently, this patient population does not have access to effective treatment within specialist healthcare services and has struggled to benefit from standard treatments. The goal of this project is to increase access to treatment tailored to their challenges. We will investigate whether a treatment program with an adapted version of Dialectical Behavior Therapy (DBT) is feasible, accepted, and perceived as useful for people with autism. The purpose of the treatment is to improve emotion regulation, function better in relationships, and avoid crises, thereby enhancing their ability to achieve personal goals, reduce suffering, and increase quality of life. Autism is a lifelong neurodevelopmental disorder, presenting with great variation and more widespread than previously thought. Difficulties with emotion regulation are a central challenge for many with autism. These difficulties often manifest as an inability to recognize, understand, and manage emotional responses, leading to destructive strategies, behaviors, and suffering. DBT is developed with a focus on emotion regulation and has shown good effects in other patient populations. The project can increase access to treatment for a patient population that currently stands without.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a lifelong neurodevelopmental condition marked by difficulties in social interaction, communication, sensory sensitivities, and repetitive behaviors. ASD varies widely among individuals and has become more recognized over time. The prevalence of ASD has significantly increased, with the U.S Centers for Disease Control and Prevention (CDC) reporting a rise from 1 in 2,222 children in 1968 to 1 in 44 children in 2020. This increase is due to evolving definitions, greater awareness, and differences in study methodologies.

Many individuals with ASD, especially those without intellectual disabilities, often remain undiagnosed until adulthood. Undiagnosed ASD is common in adult clinical populations, with a Swedish study finding that 18.9% of psychiatric outpatients had ASD. Psychiatric comorbidities are frequent in ASD, including anxiety, depression, attention deficit hyperactity disorder (ADHD), obsessive compulsive disorder (OCD), bipolar disorders, and sleep-wake disorders, complicating diagnosis and treatment. Autistic individuals often engage in suicidal behaviors, self-harm, and aggression, impacting daily life.

Autistic women without intellectual disabilities are often underdiagnosed due to less overt symptoms and their ability to camouflage difficulties. Misdiagnosis with personality disorders, particularly borderline personality disorder, is common.

Despite rising diagnosis rates, there is a lack of evidence-based treatment options for autistic adults, especially for those with comorbid mental disorders. Many clinicians lack training to work with autistic adults, and ASD specialists often lack expertise in treating co-occurring conditions. In Norway, there is a significant gap in treatment options for autistic adults without intellectual disabilities.

Emotion regulation difficulties are central challenges for many autistic adults, involving physiological arousal, brain region alterations, and unique ASD mechanisms like cognitive rigidity. Autistic adults often struggle with alexithymia, exacerbating emotion regulation issues. Developing effective emotion regulation strategies can improve quality of life.

Dialectical Behavior Therapy (DBT) helps autistic individuals manage emotions, relationships, and crises. DBT has shown effectiveness in reducing self-harm and suicidal behaviors among autistic adults. A study in North Carolina found DBT skills training feasible and acceptable for autistic adults without intellectual impairment. Similar studies have not been conducted in Nordic countries for outpatient psychiatric settings.

This study is a mixed-method feasibility study without a control group. With measurements pre and post treatment intervention. In the project period approximatly 15 patients will be invited to participate, referred to the project by a therapist form an general outpatient psychiatric clinic.

Primary objectives

If the DBT-skills training is relevant - The severity of difficulties in emotion regulation for the population, and the presences of destructive behaviour such as self-harm and suicide behaviour.

If DBT-skills training is accepted by tracking the dropout rate from DBT skills training, as well as the percentage of DBT-SUD skills sessions participated in, and the percentage completed homework.

Acceptability and Feasibility post treatment by evaluating participants' experiences with the treatment, and use of unhelpful and helpful strategies with self-rapport instruments.

Secondary objectives

Tracking the change in two target behaviors and four target emotions and use of skills in the treatment period with a diary card.

Assessing goals, hinders, and resources at the start and completion of the DBT skills training, with a qualitative interview.

Strength and limitations

Strength: This is a feasibility study in naturalistic treatment, making the results generalizable.

The result of the study gives relevant information in a population that is often excluded from studies because of ASD diagnosis.

Limitations: With a lack of a randomized control group, one cannot measure the direct effect of the intervention.

Future research: If the intervention fits the progression criteria and proves to be relevant, feasible, acceptable, and of potential benefit for the patients, the future aim is to conduct a Randomized Control Trial (RCT) on the effect of DBT skills training for autistic adults with difficulties in emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

* Fit general inclusion criteria for the out- patient treatment at the clinic.
* Have diagnosed autism, and pervasive difficulties in emotion regulation.
* Speak Scandinavian (Norwegian, Danish and/or Swedish).
* Manage to commit to participating in the DBT- skills training.
* Be willing to sign the written informed consent.

Exclusion Criteria:

* Have a clinically significant low linguistic functioning that hinders the patient in understanding and answering the questions on the self-report instruments.
* Being actively psychotic.
* Have a Body Mass Index (BMI) under 17.
* Cognitive disability Intelliganve quotient (IQ) <85

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Difficulties in emotion regulation scale (DERS) - 8 | From enrollment to the end of treatment at 28 weeks.
  a shortened self-report instrument, developed from the original DERS-36 meant to measure difficulties in emotion regulation. The DERS-8 consists of 8 items prefaced with the phrase "When I'm upset," to provide respondents with a uniform context that elicits thinking about situations requiring regulation of negative emotion; answers to items likely to represent affect, thought, and actions in response to such situations. The scale offers a brief unidimensional measure of difficulties in emotion regulation for adolescents and adults. Higher scores indicate greater levels of difficulties in emotion regulation.
participation in treatment | From enrollment to the end of treatment at 28 weeks.
  Dropout rate from DBT skills training, as well as the percentage of DBT-SUD skills sessions participated in, and the percentage completed homework.
Dialectical Behavior Therapy- Ways of Coping Checklist (DBT-WCCL) | From enrollment to the end of treatment at 28 weeks.
  It is a 59 item self-rapport questionnaire that assesses both positive and negative methods of coping with stressful situations including problem-focus, seeking social support, blaming self, blaming others, wishful thinking, and avoidance as well as DBT skills use on 4-point likert scale: 0 = Never Used, 1= Rarely Used, 2= Sometimes Used, 3 = Regularly Used. The questionnaire is divided into 2 subscales: 1) DBT skills subscale that consists of Nine items represent emotion regulation skills, seven represent interpersonal effectiveness skills, five depict mindfulness skills, 19 represent crisis survival skills, two depict reality acceptance skills (0-114). and 2) Dysfunctional Coping Subscale that consist of 17 items referring to dysfunctional behavior in general along with items referring more specifically to blaming others (0-63).

SECONDARY OUTCOMES:
Diary card | From enrollment to the end of treatment at 28 weeks.
  Tracking the change in two target behaviours and four target emotions and use of skills in the treatment period with a diary card.
Qualitative interview guide - DBT skills training ASD | From enrollment to the end of treatment at 28 weeks.
  Qualitative interview focusing on the participants goals, hinders and resources, and how they experienced the treatment interventions in relation to achieving these goals.

CONTACTS AND LOCATIONS:
Overall Officials: Egil Jonsbu, MD, PhD, Study Director — More And Romsdal Hospital Trust

REFERENCES:
- [Background] Bargiela S, Steward R, Mandy W. The Experiences of Late-diagnosed Women with Autism Spectrum Conditions: An Investigation of the Female Autism Phenotype. J Autism Dev Disord. 2016 Oct;46(10):3281-94. doi: 10.1007/s10803-016-2872-8. PMID 27457364
- [Background] Ritschel LA, Guy L, Maddox BB. A pilot study of dialectical behaviour therapy skills training for autistic adults. Behav Cogn Psychother. 2022 Mar;50(2):187-202. doi: 10.1017/S1352465821000370. Epub 2021 Sep 23. PMID 34553682

DOCUMENTS (3):
  • Study Protocol (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT07021274/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT07021274/SAP_001.pdf
  • Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT07021274/ICF_002.pdf